CLINICAL TRIAL: NCT05133804
Title: The Relation Between Attentional, Sensory and Emotional Dysregulation in Adults With Posttraumatic Stress Disorder: a Double-blind, Placebo-controlled Randomized Controlled Trial of the Combined Treatment With Reboxetine and Methylphenidate
Brief Title: Efficacy of Reboxetine and Methylphenidate Treatment on Attentional, Sensory and Emotional Dysregulation in Adults With PTSD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Haifa (Other)
Responsible Party: Principal Investigator, Avi Avital, Professor at Department of Occupational Therapy; Head of Behavioral Neurobiology lab, University of Haifa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LH9/2019
Record Dates: First submitted 2021-10-04; First posted 2021-11-24 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Posttraumatic Stress Disorder; Attention Deficit; Sensory Processing; Emotion Regulation; Methylphenidate; Reboxetine; Randomized Controlled Trial; Electroencephalogram; Functional near-infrared spectroscopy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Attention Deficit Disorder with Hyperactivity; Emotional Regulation | interventions — Methylphenidate; Reboxetine

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into two groups: either treatment with medication or treatment with placebo.
  In addition, within each group patients will be randomized into a group for EEG recording and a group for fNIRS recording. This is a non-interventional randomization.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment with Reboxetine and Methylphenidate (Experimental): During the first 3 weeks of the study, subjects in the active treatment group will take reboxetine at a dose of 4mgper day, with the instructions to start at 2mg per day for 3 days and then increase the dosage to 4mg per day for 26 days, i.e. until completion of the study.
  On day 22 of the study, the patients will take the first dosage of10mg Ritalin or a placebo, and remain in the clinic for 2 hours to guard safety and guidance during possible occurrence of side effects such as anxiety, palpitations, etc. During the observation time in the clinic, 6 Ritalin IR 10mg and 3 Reboxetine 4mg pills will be handed out to the participants. These pills will be taken at the responsibility of the subject at8:00 AM (Ritalin and Reboxetine) and at noon (Ritalin only) at the following three days.
  Interventions: Drug: Methylphenidate; Drug: Reboxetine
- Treatment with Placebo (Placebo Comparator): The patients will take placebos according to the medication schedule of the treatment group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylphenidate — Ritalin 10mg
  Other Names: Ritalin
  Arms: Treatment with Reboxetine and Methylphenidate
Drug: Reboxetine — Reboxetine 4mg
  Arms: Treatment with Reboxetine and Methylphenidate
Drug: Placebo — Placebo matched to Reboxetine
  Other Names: Placebo matched to Reboxetine
  Arms: Treatment with Placebo
Drug: Placebo — Placebo matched to Ritalin
  Other Names: Placebo matched to Ritalin
  Arms: Treatment with Placebo

SUMMARY:
Up-to-date, no studies have examined the attentional, sensory and emotional processing (difficulties) among patients diagnosed with Posttraumatic Stress Disorder (PTSD). In addition, the efficiency of drug treatments that focus on the noradrenergic and dopaminergic, and thus influence attention processing and PTSD symptoms through these pathways, have only briefly been investigated. There is well-established and long-standing evidence for the involvement of dopamine and noradrenaline in attentional function. This previously led to an investigation by the investigator's research lab in which the investigators hypothesized the involvement of an attentional disorder would influence PTSD symptoms in a rat model. Based on these results, the current study aims to characterize attentional deficits in patients with PTSD, as well as the correlation between attention, emotional regulation and sensory processing. The investigators do this partially by conducting a case-control study and through a subsequent double-blind RCT (with only the cases). The patients will be either treated with reboxetine + methylphenidate or placebo.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is a highly impairing psychiatric disorder, characterized by re-experiencing, avoidance behaviour, emotional numbing, and hyperarousal after traumatic exposure. Current treatments mainly focus on non-cognitive symptoms and are only partially effective: one third of PTSD patients will find symptoms to be chronic and progressive; highly impacting daily function and quality of life. Arising evidence suggests a correlation between impaired attention, sensory dysfunction, and PTSD symptoms. Thus, the importance of combined treatment, focused on concentration difficulties as often found PTSD, has been suggested. Two suggested leads are reboxetine and methylphenidate.

Hypothesising that impaired attentional and sensory processing induces re-experiencing with avoidance and hyperarousal as coping strategies, the investigators aim to elucidate the neuro-dysregulation characteristics of each of the PTSD symptoms, with focus on attention, executive function and sensory processing, and relate to their implications on daily life function, following a novel combined treatment strategy of reboxetine and methylphenidate (Ritalin).

A case-control study will be conducted, including 53adult patients with PTSD and 53 matched healthy controls. First, a baseline measure will be performed amongst all participants to create a population profile. Then, patients will be randomised into an active treatment group (n=27) and a placebo group (n=26) for a double-blind randomized controlled trial, investigating the effect of a 3-week treatment with reboxetine 4mg per day and a one-week addition of Ritalin 10mg twice a day.

This research will include established and innovative neurophysiological measures and questionnaires. A PTSD symptom profile will be created combining the Clinician-Administered Posttraumatic Stress Disorder Scale and Posttraumatic Stress Disorder Symptom Scale. Brain activity will be measured using functional near-infrared spectroscopy (fNIR) or electroencephalography, with the Auditory Sustained Attention Test (ASAT) and Electrodermal Activity (EDA). Together with the Conners' Adult Attention Deficit Hyperactivity Disorder (ADHD) Rating Scale - Short Version, the ASAT and EDA will create an attentional profile. Furthermore, a sensory profile consisting of the Adolescent/Adult Sensory Profile Questionnaire, and an executive function profile measured with the Behavior Rating Inventory of Executive Function will be created. Finally, in order to relate to individual experiences in real-life context, this research measures activities through the Daily Living Questionnaire and quality of life with the World Health Organization Quality of Life Instrument.

Using a translational research paradigm, this research is one of the first to investigate neuro-dysregulation in PTSD with a focus on sensory processing and executive function, with emphasis on attention and behaviour. It is also the first research to integrate the fNIR with the ASAT and EDA, thus contributing to the technological advancing of clinical research. This research will gather innovative data that may offer new explanations of PTSD symptoms and allow for further development of treatment interventions needed to reduce the burden of disease and optimise quality of life.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with PTSD according to DSM-IV or DSM-5 criteria
* current treatment at the outpatient facilities of Lev HaSharon Netanya Adult Clin
* age between 20 and 60 years
* PTSD diagnosis at least one month prior to study inclusion
* no present-day re-exposure to the traumatic event
* any psychotropic drug therapy that is being administered must be at a fixed dose for at least one month prior to the study conductance

Exclusion Criteria:

1. comorbid major psychiatric disorder, e.g. psychotic disorder, unipolar or bipolar disorder, borderline personality disorder, or active suicidal ideation,
2. ADHD diagnosis,
3. significant or severe systematic disease that limits normal activity, e.g. autoimmune disease, AIDS or renal failure,
4. cardiovascular disease, e.g. hypertension, atrioventricular (AV) block, bradycardia, or conduction disorder,
5. severe disease that is a threat to life, e.g. acute myocardial infarction, respiratory failure, or cancer,
6. nervous system impairment, e.g. multiple sclerosis, Alzheimer's disease, Parkinson's disease, epilepsy, or stroke,
7. previous or current severe traumatic brain injury,
8. glaucoma,
9. impaired hearing,
10. pregnancy or breastfeeding during study inclusion,
11. active substance dependency including regular use of medical cannabis,
12. use of steroid medication in the two months prior to study conductance,
13. use of medication that may affect the function of the central nervous system,
14. failure to complete all research steps

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Clinician-Administered Posttraumatic Stress Disorder Scale for the Diagnostic and Statistical Manual (DSM)-5 (CAPS-5) between baseline score (before treatment) and score on day 26 (after treatment) | Day 1 and day 26
  PTSD symptom severity score. Total of 56 questions. Minimum score 0, maximum score 80. A higher score reflects a worse outcome.

SECONDARY OUTCOMES:
Posttraumatic Stress Disorder Symptom Scale (PSS-SR5) | Day 1 and day 26
  PTSD symptom severity score. Total of 24 questions. Minimum score 0, maximum score 80. A higher score reflects a worse outcome.
Conner's Adult ADHD Rating Scales - Self Report: short version (CAARS-S:S) | Day 1 and day 26
  ADHD index score. Total of 26 questions. Minimum score 26, maximum score 78. A higher score reflects a worse outcome.
Electroencephalography (EEG) | Day 1, day 21 and day 26
  Electrical brain activity, measured through event-related potentials (ERP)
Functional near-infrared spectroscopy (fNIRS) | Day 1, day 21 and day 26
  Cortical hemodynamic activity, measured through concentrations of oxygenated and deoxygenated hemoglobin.
Electrodermal Activity (EDA) | Day 1, day 21 and day 26
  Electrodermal activity, measured through sweat secretion on digit 2 and digit 4 of right hand.
Auditory Sustained Attention Test (ASAT) | Day 1, day 21 and day 26
  Pre-pulse inhibition, measured through the eyeblink reflex at the level of the musculus orbicularis oculi 1cm below the pupil.
Adolescent/Adult Sensory Profile Questionnaire (AASP) | Day 1 and day 26
  Sensory profile. Total of 60 questions. Minimum score 60, maximum score 300. A higher score reflects a worse outcome.
Behavior Rating Inventory of Executive Function - Adult Version (BRIEF-A) | Day 1 and day 26
  Global executive composite. Total of 75 questions. Minimum score 75, maximum score 225. A higher score reflects a worse outcome.
Daily Life Questionnaire (DLQ) | Day 1 and day 26
  Daily life limitations. Total of 59 questions. Minimum score 28, maximum score 112. A higher score reflects a worse outcome.
World Health Organization Quality of Life Questionnaire - BREF (WHOQOL-BREF) | Day 1 and day 26
  Quality of Life. Total of 26 questions. Minimum score 24, maximum score 120. A higher score reflects a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Avi Avital, PhD, Principal Investigator — University of Haifa; Batya Engel-Yeger, PhD, Principal Investigator — University of Haifa; Inbal Brenner, MD, Principal Investigator — Lev HaSharon Mental Health Center; Tsipi Milman, MD, Principal Investigator — Emek Medical Center
Locations (3):
- Israel (3):
  - Emek Medical Center, Afula
  - University of Haifa, Haifa
  - Lev HaSharon Mental Health Center, Netanya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aga-Mizrachi S, Cymerblit-Sabba A, Gurman O, Balan A, Shwam G, Deshe R, Miller L, Gorodetsky N, Heinrich N, Tzezana O, Zubedat S, Grinstein D, Avital A. Methylphenidate and desipramine combined treatment improves PTSD symptomatology in a rat model. Transl Psychiatry. 2014 Sep 23;4(9):e447. doi: 10.1038/tp.2014.82. PMID 25247592
- [Background] McAllister TW, Zafonte R, Jain S, Flashman LA, George MS, Grant GA, He F, Lohr JB, Andaluz N, Summerall L, Paulus MP, Raman R, Stein MB. Randomized Placebo-Controlled Trial of Methylphenidate or Galantamine for Persistent Emotional and Cognitive Symptoms Associated with PTSD and/or Traumatic Brain Injury. Neuropsychopharmacology. 2016 Apr;41(5):1191-8. doi: 10.1038/npp.2015.282. Epub 2015 Sep 11. PMID 26361060